CLINICAL TRIAL: NCT00736931
Title: Randomized, Comparative, Double-blind, Placebo-controlled, Triple-dummy, Four-way Cross-over Study to Investigate Neurocognitive Effects of Brivaracetam in Healthy Subjects
Brief Title: Clinical Study in Healthy Volunteers to Investigate the Neurocognitive Effects of a New Antiepileptic Drug: Brivaracetam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N01297
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2008-10

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Cognitive neurophysiological tests (CNT); Neuropsychological assessments
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam; Levetiracetam; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 4 arms (in cross-over): brivaracetam, levetiracetam, lorazepam and placebo.
  Interventions: Drug: Brivaracetam
- 2 (Active Comparator): 4 arms (in cross-over): brivaracetam, levetiracetam, lorazepam and placebo.
  Interventions: Drug: levetiracetam
- 3 (Active Comparator): 4 arms (in cross-over): brivaracetam, levetiracetam, lorazepam and placebo.
  Interventions: Drug: lorazepam
- 4 (Placebo Comparator): 4 arms (in cross-over): brivaracetam, levetiracetam, lorazepam and placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Brivaracetam — Brivaracetam 10 mg tablets
  Arms: 1
Drug: levetiracetam — 500mg tablets
  Arms: 2
Drug: lorazepam — lorazepam 2 mg over encapsulated tablets
  Arms: 3
Other: placebo — placebo capsules
  Arms: 4

SUMMARY:
The primary objective of the study is to evaluate the neurocognitive effects of brivaracetam

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer aged 18 to 50 years inclusive
* Body Mass Index (BMI) between 18.0 and 30.0 kg/m² inclusive
* Good physical and mental health status
* Blood pressure and heart rate within normal range
* Electrocardiogram and laboratory tests without clinically significant abnormality

Exclusion Criteria:

* IQ ≤ 80 as determined by Test of non-verbal intelligence
* Center for Epidemiological Studies Depression (CES-D Scale ≥16,
* Known allergy/intolerance to pyrrolidinone derivatives
* Abnormalities on EEG recordings
* Pregnant, lactating women
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, neurological, psychiatric disorders
* Use of any hepatic enzyme-inducing drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Summary score from a Cognitive Neurophysiological Test (derived from electroencephalogram [EEG], event related potentials [ERP], and cognitive performance measures) | 3 weeks

SECONDARY OUTCOMES:
Component subscores from the Cognitive Neurophysiological Test and scores from neuropsychological tests/assessments: SSEQ Subject Self Evaluation Questionnaire. SMDT Symbol Digit Modalities Test. COWA Controlled Oral Word Association. MCG Parag | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Overland Park, Kansas, United States

REFERENCES:
- [Derived] Meador KJ, Gevins A, Leese PT, Otoul C, Loring DW. Neurocognitive effects of brivaracetam, levetiracetam, and lorazepam. Epilepsia. 2011 Feb;52(2):264-72. doi: 10.1111/j.1528-1167.2010.02746.x. Epub 2010 Sep 30. PMID 20887370